CLINICAL TRIAL: NCT01103765
Title: A Prospective Randomized Multicenter Study of the Efficacy and Safety of Systematic Post -Dilatation With Noncompliant Balloon After Successful Drug-eluting Stent Implantation. IVUS Analysis.
Brief Title: Post-dilatation for Optimization of Drug-eluting Stents (DES) Deployment Assessed by Intravascular Ultrasound Multicenter Analysis
Acronym: PODIUM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Recherches et etudes en sciences sociales et sante, France (Network)
Responsible Party: Dr Georgios SIDERIS, Assistance Publique - Hôpitaux de Paris
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UK0801
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Implant
Keywords: Post-dilatation; noncompliant balloon; optimal stent deployment of drug-eluting stent; Intravascular ultrasound (IVUS); Optimal stent deployment defined by intravascular ultrasound analysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- classic strategy (Placebo Comparator): after drug-eluting stent(DES) deployment perform of Intravascular ultrasound analysis without post-dilatation
  Interventions: Procedure: stent deployment without post-dilatation
- post-dilatation strategy (Active Comparator): After drug-eluting stent (DES) deployment IVUS analysis and systematic post-dilatation with noncompliant balloon 0.25mm larger than stent balloon. After post dilatation new IVUS analysis.
  Interventions: Procedure: post dilatation after stent deployment

INTERVENTIONS:
Procedure: post dilatation after stent deployment — Post-dilatation with a noncompliant balloon larger 0.25mm than stent balloon.
  Arms: post-dilatation strategy
Procedure: stent deployment without post-dilatation — stent deployment without systematic post dilatation
  Arms: classic strategy

SUMMARY:
Comparison with use of Intravascular Ultrasound (IVUS) analysis of two methods of percutaneous coronary interventions (PCI) with drug eluting stent:

After successful drug eluting stent implantation, patients were randomized into two groups: Group A had no further dilatation, and Group B had additional post-dilatation with a noncompliant balloon. The investigators performed IVUS analysis in groups A and B just before randomization and after post-dilatation in group B.

DETAILED DESCRIPTION:
Stent expansion of DES using current stent deliver systems is frequently suboptimal. Further more smaller minimal stent area (MSA) and stent underexpansion following deployment of DES are strong predictors of stent thrombosis and (TVR) target vessel revascularization. The investigators hypothesize than adjunctive postdilatation with noncompliant balloon can improve DES deployment.

After successful drug eluting stent implantation, patients will be randomized into two groups: Group A with no further dilatation, and Group B with additional post-dilatation with a noncompliant balloon. The investigators will performed IVUS analysis in groups A and B just before randomization and after post-dilatation in group B. Post dilatation will be performed with noncompliant balloon and with a nominal diameter 0.25mm larger than stent balloon.

The primary endpoint is optimum stent deployment. For defining the optimal stent deployment the investigators use the IVUS criteria adopted in the MUSIC study: Complete apposition without underexpansion and with symmetric stent expansion.

Patients are eligible after successful drug-eluting stent implantation in a native coronary artery. Patients with myocardial infarction or acute coronary syndrome will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Successful drug eluting stent implantation in a native coronary artery

Exclusion Criteria:

* Percutaneous coronary intervention (PCI) of Left main coronary artery;
* Myocardial infarction;
* Acute coronary syndrome;
* Emergency PCI;
* PCI for in-stent restenosis;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Optimal stent deployment defined by IVUS analysis | at 18 months
  The primary endpoint is optimum stent deployment. For defining the optimal stent deployment we use the IVUS criteria adopted in the MUSIC study: Complete apposition without underexpansion and with symmetric stent expansion. All patients(group A and B) will have IVUS analysis for defining optimal stent deployment

SECONDARY OUTCOMES:
Complications of percutaneous coronary intervention (PCI) | at day0, at day1, at the end of hospitalisation and year1
  Death,Myocardial infarction, coronary dissection, intracoronary thrombosis, target vessel revascularisation.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios SIDERIS, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de cardiologie interventionnelle - Hôpital Lariboisière, Paris, France